CLINICAL TRIAL: NCT01473693
Title: Changes in Brain Structure Related to Systemic Chemotherapy Treatment: A Prospective Study in Individuals Diagnosed With Non-small Cell Lung Cancer Utilizing High-resolution Structural Magnetic Resonance Imaging
Status: Terminated | Type: Observational
Why Stopped: Lack of Accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-145
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Quality of Life; Lung cancer; MRI; Surgery; induction chemotherapy; 11-145
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy; Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- surgery-only group: This will be a prospective study to investigate chemotherapy related structural brain changes in individuals undergoing anatomic lung resection for non-small cell carcinoma with and without, induction systemic chemotherapy treatment.
  Interventions: Other: MRI Screening Form, MRI, Demographic / Medical Data form
- induction chemotherapy group: This will be a prospective study to investigate chemotherapy related structural brain changes in individuals undergoing anatomic lung resection for non-small cell carcinoma with and without induction systemic chemotherapy treatment.
  Interventions: Other: MRI Screening Form, MRI. Demographic / Medical Data

INTERVENTIONS:
Other: MRI Screening Form, MRI, Demographic / Medical Data form — MRI Screening Form: MRI screening form will be administered twice at baseline and follow up visits. Administration time: 5 minutes. MRI data: at both time points (pre- and post-treatment only) Administration time: 30 minutes.
  Demographic / Medical Data: Administration time: 5 minutes.
  Groups: surgery-only group
Other: MRI Screening Form, MRI. Demographic / Medical Data — MRI Screening Form: MRI screening form will be administered twice at baseline and follow up visits Administration time: 5 minutes.
  MRI data: at both time points (pre- and post-treatment only) Administration time: 30 minutes.
  Demographic / Medical Data: Administration time: 5 minutes
  Groups: induction chemotherapy group

SUMMARY:
The purpose of this study is to learn about the effects of cancer treatment on the brain. Some cancer patients report changes in their memory or thinking after treatment. These changes could be a result of changes in brain structure, such as a change in size or thickness of different parts of the brain. The investigators will look to see if these changes in brain structure happen through the results of magnetic resonance imaging (MRI). The investigators will do this by looking at the brain structure of lung cancer patients who have surgery and chemotherapy versus those who have surgery only.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 years old
* As per self report and/or medical record female patients are either postmenopausal or not able to become pregnant
* Patients with biopsy proven or suspected non-small cell lung cancer planned to undergo induction chemotherapy and surgery, OR with biopsy proven or suspected non-small cell lung cancer planned to undergo immediate surgical resection
* No clinical/neurological symptoms suggestive of brain metastases by attending's judgment as documented in the medical record and/or correspondence with the research team
* In the judgement of the consenting professional, patient is able to understand English, through verbal and written communication
* Patient is able to undergo MRI scanning (verified with pre-MRI Safety Screening form (Appendix A) used in MSKCC MRI Centers) completed at screening and again prior to having the MRI.

Exclusion Criteria:

* Patients with history of significant neurological diagnoses including stroke, tumor, dementia, epilepsy, or multiple sclerosis as indicated by medical records and/or self report
* History of head injury with evidence of brain injury or loss of consciousness for > 60 minutes as per EMR or self-report
* No prior treatment with chemotherapy
* Participant has dentures, body jewelry or wig that they are unable to remove as per self-report
* Patient reports that he/she cannot undergo MRI scanning without significant distress or discomfort
* Significant psychiatric or cognitive disturbance sufficient, in the investigator's judgment, to preclude providing informed consent or participating in the study (i.e., schizophrenia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic Oncology, Radiation Oncology, Surgery or Ambulatory Care clinic lists
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
longitudinal structural changes in the brain | 1 month following completion of a 6 month course of induction chemotherapy or 7 months following surgery
  Using MRI in patients diagnosed with non-small cell lung cancer in either the induction chemotherapy exposed or surgery-only group in dorsolateral prefrontal cortex or bilateral hippocampus

SECONDARY OUTCOMES:
longitudinal structural changes in the brain | 1 month following completion of a 6 month course of induction chemotherapy
  Using MRI in patients diagnosed with non-small cell lung cancer in the induction chemotherapy exposed group in dorsolateral prefrontal cortex or bilateral hippocampus.

CONTACTS AND LOCATIONS:
Overall Officials: James C Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm